CLINICAL TRIAL: NCT00224263
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Assess the Efficacy and Safety of Lingzhi in Patients With Early Parkinson's Disease Receiving Stable L-dopa/DCI
Brief Title: Efficacy and Safety of Lingzhi in Patients With Early Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004BA702B02
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Parkinson's Disease
Keywords: Traditional Chinese Medicine; Lingzhi
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lingzhi (Ganoderma)

SUMMARY:
The purpose of this study is to determine whether Lingzhi (Ganoderma), a widely used traditional Chinese Medicine is effective and safe in the treatment of Parkinson's disease when combined use with L-dopa.

DETAILED DESCRIPTION:
This study is to focus on the effects of Lingzhi on non-motor symptoms of Parkinson's diseases as the primary outcome and on delaying the disease progression using the delay start design as the secondary outcome measurement. Two dosage groups and one placebo control group with total 360 subjects will be recruited. The treatment is one year.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give informed consent
* age 30 years or older at time of diagnosis of Parkinson's disease
* have idiopathic Parkinson's disease, defined as:

  * having at least 2 of the following 4 signs: resting tremor, bradykinesia, rigidity, or postural reflex impairment, at least one of which must be resting tremor or bradykinesia
  * no secondary or atypical parkinsonism
  * asymmetric features (current signs or history of asymmetric onset)
  * response to L-dopa, by patient self-report
* Parkinson's disease duration of no more than 5 years
* receiving stable therapy of L-dopa/DCI for at least 3 months; acceptable dose range: 250 mg - 1000 mg L-dopa/DCI daily
* Hoehn and Yahr stage < 4 on stable L-dopa/DCI treatment

Exclusion Criteria:

* have atypical parkinsonism due to drugs, metabolic disorders, encephalitis, or other neurodegenerative diseases
* have any other known medical or psychiatric condition that may compromise their participation in the study
* have taken another investigational drug within 90 days of baseline
* have a change in dosage of any other antiparkinsonian drug (eg, pramipexole, ropinirole, pergolide, bromocriptine, methylphenidate, anticholinergics, or amantadine) during the study or within 90 days prior to baseline
* have received treatment with dopamine blocking agents (including neuroleptic agents, antiemetic agents), dopamine-depleting agents (including reserpine or tetrabenazine) within 90 days prior to baseline
* do not consent to participate

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2005-09; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Motor Function

SECONDARY OUTCOMES:
Cognition
Mood
Quality of Daily Life

CONTACTS AND LOCATIONS:
Overall Officials: Piu Chan, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China